CLINICAL TRIAL: NCT02958553
Title: EmPOWERing Active Seniors With Energy
Acronym: EASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Collaborators: BionX Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P16-01
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Amputation
Keywords: Lower Extremity Limb Loss; Prosthesis Use

STUDY DESIGN:
Intervention Model Description: First the patient data is gathered with the subject's own passive prosthetic. Then switched over to the emPOWER Ankle. Third, the patient's prosthetic is switched back to test for carry-over benefits. Then they are put on the emPOWER for a final series of tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- emPOWER Ankle (powered prosthesis) (Other): The subject's own passive prosthesis will be used as a baseline and crossed over after the emPOWER has been worn 3-4 months. Then the passive foot will be crossed back to the emPOWER for a final series of tests.
  Interventions: Device: emPOWER Ankle; Device: Subject's own passive prosthesis

INTERVENTIONS:
Device: emPOWER Ankle — The device is 510k cleared and is intended to replace a missing foot and ankle. The emPOWER Ankle is to be used exclusively for fittings of lower-extremity amputations as prescribed by a healthcare professional.
Device: Subject's own passive prosthesis — Devices will vary. Data gathered will form a baseline.

SUMMARY:
A pilot study comparing the emPOWER Ankle System to standard carbon fiber prosthetic feet, in active seniors.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the increase in the distance subjects can walk during a six (6) minute period while wearing the emPOWER Ankle compared to a passive lower-extremity prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 55 years or older
* Subjects with transtibial amputations of either leg at least 1 year prior
* Suction or elevated vacuum suspension and Socket Comfort Score of at least 6
* Sock fluctuation of ≤ 8 ply per day
* K-level rating of 3 or 4 based on the Amputee Mobility Predictor Assessment Tool
* Ability to walk at a walking speed of > 0.75 meters per second
* Unilateral amputees (up to 7 bilateral amputees can be included, 1 per site in addition to the unilateral amputees who will be analyzed as a separate sub group)
* Foot size: 25-30 cm
* Ability to complete a continuous 6-Minute Walk Test
* Ability to provide written, informed consent
* Ability to complete study visits and study documents
* Ability to manage the complexity of a powered device including charging and changing batteries as needed
* Ability to read and understand English

Exclusion Criteria:

* Subjects who have never used a prosthetic device
* Less than 55 years of age
* Weight <150 lbs. or > 287 lbs.
* Transfemoral amputees
* Active sores or ulceration on subject's residual limb
* Sore on contralateral foot.
* Cuff-link socket suspension
* Socket Comfort Score less than 6
* Sock fluctuation of > 8 per day
* K level of 1 or 2
* Amputation clearance < 8.625"
* History of stroke or TIA that impairs current walking
* Recent history of excessive falling defined as more than 2 falls requiring medical assistance in the prior year
* Medications potentially affecting balance
* Recent hospitalization (within past 3 months)
* Cognitive deficiency that would impact ability to charge and change batteries as needed

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Melton, M.D., Principal Investigator — Principal Investigator
Locations (1):
- UTHealth, Department of Orthopedic Surgery, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The EmPOWERing Active Seniors with Energy Study first subject was enrolled February 10, 2017. The last subject was enrolled November 6, 2017. All subjects were enrolled at a single study site which was a lower-limb rehabilitation clinic.
Period: Phase I, 1st Visit -Passive Prosthesis
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 8
Completed | 8
Not Completed | 0
Period: Phase I, 2nd Visit -Fitted With emPOWER
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 8
Completed | 8
Not Completed | 0
Period: Phase I, 3rd Visit -2 Week emPOWER FU
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Phase II, 4th Visit -3 Month emPOWER FU
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 7 (Only 4 subjects started Phase II of the study. Phase II was optional per protocol.)
Completed | 4
Not Completed | 3
Period: Phase II, 5th Visit -Crossover Visit
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 4
Completed | 4
Not Completed | 0
Period: Phase II, 6th Visit -6 Month emPOWER FU
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 2
Period: Phase II, 7th Visit -12 Month emPOWER FU
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 8 patients completed Visit 1 and have Baseline information available
Groups:
- emPOWER Ankle (Powered Prosthesis): The subject's own passive prothesis will be used as a baseline and crossed over after the emPOWER has been worn for 3-4 months. Then the passive foot will be crossed back to the emPOWER for a final series of tests.
  emPOWER Ankle: The deivce is 510k cleared and is intended to replace a missing foot and ankle. The emPOWER ankle is to be used exclusively for fittings of lower-extremity amputations as prescribed by a healthcare professional.
  Subject's own passive prosthesis: Devices will vary. Data gathered will form a baseline.
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Six Minute Walk Test (6MWT)
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in the walking distance measured by the Six Minute Walk Test (6MWT). 6minWT improvement was defined as a minimum increase of 45 meters.
Time Frame: 3 months with the emPOWER ankle
Population: The results for the primary effectiveness endpoint for improvement in walking distance with the Empower compared to the distance walked with the subject's passive prosthesis as measured by the 6 minute Walk Test (6MWT) at 3 months from four subjects were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

2. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Twelve Minute Walk Test (12MWT)
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in the walking distance measured by the Twelve Minute Walk Test (12MWT). 12minWT improvement was defined as a minimum increase of 90 meters.
Time Frame: 3 months with the emPOWER ankle
Population: The results for the secondary effectiveness endpoint for improvement in walking time with the Empower compared to the distance walked with the subject's passive prosthesis as measured by the 12 minute Walk Test (12MWT) at 3 months from four subjects were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 2
  No Change | 2
  Declined | 0

3. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the 10 Meter Walk Test (10MWT)
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in the walking distance measured by the 10 Meter Walk Test (10MWT). 10MWT improvement was defined as a minimum increase of 0.1 m/s.
Time Frame: 3 months with the emPOWER ankle
Population: The results for the secondary effectiveness endpoint for improvement in walking distance with the Empower compared to the distance walked with the subject's passive prosthesis as measured by the 10MWT at 3 months from four subjects were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

4. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the L-Test
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in the walking time measured in the L-Test. L-Test improvement was defined as a minimum decrease of 4.5 seconds.
Time Frame: 3 months with the emPOWER ankle
Population: The results for the secondary effectiveness endpoint for improvement in walking distance with the Empower compared to the distance walked with the subject's passive prosthesis as measured by the L-Test at 3 months from four subjects were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 0
  No Change | 4
  Declined | 0

5. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Ramp Test
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in the walking time measured in theRamp Test. Ramp Test improvement was defined as a minimum decrease of 6 seconds to complete the test.
Time Frame: 3 months with the emPOWER ankle
Population: The results for the secondary effectiveness endpoint for improvement in walking distance with the Empower compared to the distance walked with the subject's passive prosthesis as measured by the Ramp Test at 3 months from four subjects were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 0
  No Change | 2
  Declined | 2

6. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Activities-specific Balance Confidence (ABC) Scale Score
Description: The proportion of patients with a clinically meaningful change (improvement, no change, worsening) in abulatory activities measured by the Activities-specific Balance Confidence Scale. Improvement in the ABC was defined as a minimum detectable change of 13% increase in score.
  The ABC Scale is a self-administered questionnaire that asks the patient to rate his or her confidence in performing various ambulatory activities on a scale from 0% (no confidence) to 100% (complete confidence) without losing balance or becoming unsteady. Scores for each of the 16 items will be collected and an average percentage calculated, with scores <67 indicating an increased risk of falling.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in ABC scale with the Empower at 3 months compared to the ABC scale with the subject's passive prosthesis as measured by the ABC scale.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

7. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Falls Efficacy Scale Score
Description: The Falls Efficacy Scale is a validated 10-item self-report questionnaire designed to assess confidence in the ability to perform 10 activities of daily living without falling as an indicator of how one's fear of falling impacts physical performance. Each item is rated from 1 ("very confident") to 10 ("not confident at all"), and the per item ratings are added to generate a summary total score (10 to 100). Lower scores indicate more confidence and higher scores indicate lack of confidence and greater fear of falling. It has been validated for use in the elderly and persons with amputations. Scores ≥70 indicate an increased fear of falling. Improvement in the Falls Efficiacy Scale was defined as a minimum increase of 2 in the score.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in Falls Efficiacy scale with the Empower at 3 months compared to the Falls Efficiacy scale with the subject's passive prosthesis as measured by the Falls Efficiacy scale.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Improvement | 3
  Declined | 0

8. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Amputee Mobility Predictor (AMP) Assessment
Description: The AMP is an instrument designed to measure ambulatory potential of lower-limb amputees. Subjects begin the test seated in a hard chair with arms and are tested for a total of 21 items assessing abilities of increasing level of difficulty. Abilities assessed include sitting balance, transfer from chair to chair, standing balance, gait quality, negotiating obstacles, and the use of assistive devices. The total score range for the AMP is 0 to 47 points. A minimal detectable change of 4 points was the definition of improvement.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in AMP with the Empower at 3 months compared to the AMP with the subject's passive prosthesis as measured by the AMP Assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 0
  No Change | 4
  Declined | 0

9. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Prosthetic Limb Users Survey of Mobility PLUS-M (12 Item Short Form)
Description: The PLUS-M is a valid and reliable self-reported measure for the mobility of adults with lower limb amputations. PLUS-M asks about the patient's ability to perform simple and complex tasks. High PLUS-M scores correspond with greater mobility. Improvement in the Mobility PLUS-M (12 item Short Form) was defined by a minimum detectable change of an increase of 5 points in the total score.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in PLUS-M with the Empower at 3 months compared to the PLUS-M with the subject's passive prosthesis as measured by the PLUS-M measure.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

10. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Patient Specific Functional Scale (PSFS)
Description: The PSFS is a self-report, goal-attainment measure aimed at identifying functional status limitations that are most relevant to individual patients. The PSFS is a reliable, valid, and efficient measure for detecting clinical change in persons with low back pain and knee dysfunction. Subjects were asked to identify three to five activities that they are having difficulty or are unable to perform because of their injury/condition. For the specified activities, patients were asked to rate their ability to perform each activity at that time (0-10 numerical scale) with '0' being unable to perform the activity, and '10' being able to perform the activity at the same level as they could prior to the injury/condition. The total score was calculated as the sum of the activity scores divided by the number of activities. Changes of >2 in the total score compared to baseline were considered "Improved."
Time Frame: 3 months with the emPOWER ankle
Population: While 4 subjects completed the PSFS, the results from only one subject were available for analysis, since 3 subjects rated different goals at each time point. The secondary effectiveness endpoint was improvement in PSFS with the Empower at 3 months compared to the PSFS with the subject's passive prosthesis as measured by the PSFS.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 1
Participants
  Improved | 1
  No Change | 0
  Worsened | 0

11. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in the Numeric Pain Rating Scale (NPRS)
Description: The NPRS is a valid and reliable measure of pain that may be used across all musculoskeletal injuries/conditions and complements the PSFS. The patient was asked to rate the pain of their joints, foot, lower back, and if they are using an assistive device any additional affected limbs on average over the last 24 hours on a scale 1-10, with '1' being 'very mild' and '10' being the 'unimaginable unspeakable'. The scores on the NPRS instruments with the emPOWER Ankle were compared to the scores on the subject's passive prosthesis. An improvement was considered a positive change of 1 for at least one area without a corresponding decrease in another.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in NPRS with the Empower at 3 months compared to the NPRS with the subject's passive prosthesis as measured by the NPRS.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 2
  No Change | 1
  Declined | 1

12. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in Activity (Monitoring Using a Fitbit Over 2-week Periods)
Description: A Fitbit activity monitor was worn to record the number of steps the Subject took with the prosthesis. The patient returned to the site with the activity monitor and the steps counted were downloaded from the device. In addition, the Subjects were sent home with a prepaid envelope and instructed to mail back the activity monitor if the next visit was more than 3 weeks later, to ensure that the data was not lost. The step counts were downloaded from the device the day the activity monitor was returned to the Investigator. The Investigator recorded the date the patient was affixed with the activity monitor, the date they received the returned activity monitor, and the date they synced the monitor. An improvement was defined as an increase in the average daily step count of 750 steps.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in activity with the Empower at 3 months compared to the activity with the subject's passive prosthesis as measured by the steps counts from the Fitbit Activity Monitor.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 3
Participants
  Improved | 0
  No Change | 1
  Declined | 2

13. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in PROMIS Physical Function
Description: PROMIS item banks and their short forms are a reliable and precise measurements of patient reported outcome measures. The scores on the PROMIS instruments with the emPOWER Ankle 3 months after fitting will be compared to the scores on the subject's passive prosthesis. PROMIS Physical Function improvement was defined as a minimally clinically important difference (MCID) of an increase of 6.8 in a total score.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in PROMIS Physical Function with the Empower at 3 months compared to PROMIS Physical Function with the subject's passive prosthesis as measured by the PROMIS Physical Function.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 2
  No Change | 2
  Declined | 0

14. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in PROMIS Global Health Short Form
Description: PROMIS item banks and their short forms are a reliable and precise measurements of patient reported outcome measures. The scores on the PROMIS instruments with the emPOWER Ankle 3 months after fitting will be compared to the scores on the subject's passive prosthesis. PROMIS Global Health Short Form improvement was defined as an increase in a total score of 3.5.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in PROMIS Global Health with the Empower at 3 months compared to PROMIS Global Health with the subject's passive prosthesis as measured by the PROMIS Global Health Short Form.
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

15. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in PROMIS Fatigue Short Form (7a)
Description: PROMIS item banks and their short forms are a reliable and precise measurements of patient reported outcome measures. The scores on the PROMIS instruments with the emPOWER Ankle 3 months after fitting will be compared to the scores on the subject's passive prosthesis. PROMIS Fatigue Short Form (7a) improvement was defined as a minimally clinically important difference (MCID) of an increase of 5 in a total score.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in PROMIS Fatigue with the Empower at 3 months compared to PROMIS Fatigue with the subject's passive prosthesis as measured by the PROMIS Fatigue Short Form (7a).
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

16. Secondary Outcome: Number of Participants With Improvement, No Change, or Worsening in Performance in PROMIS Pain Intensity Short Form (3a)
Description: PROMIS item banks and their short forms are a reliable and precise measurements of patient reported outcome measures. The scores on the PROMIS instruments with the emPOWER Ankle 3 months after fitting will be compared to the scores on the subject's passive prosthesis. PROMIS Pain Intensity Short Form (3a) improvement was defined as a minimally clinically important difference (MCID) of an increase of 6.9 in a total score.
Time Frame: 3 months with the emPOWER ankle
Population: The results from four subjects were available for analysis for the secondary effectiveness endpoint for improvement in Pain Intensity with the Empower at 3 months compared to Pain Intensity with the subject's passive prosthesis as measured by the Pain Intensity Short Form (3a).
Measure: Count of Participants; unit: Participants
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 4
Participants
  Improved | 1
  No Change | 3
  Declined | 0

17. Other Pre Specified Outcome: Activity Diary
Description: Self-Report Diary: Falls and daily activity. This was used to capture daily step counts from the Fitbit, daily activity and adverse events. It was a data collection tool, but was originally named as an Secondary Outcome.
Time Frame: 3 months
Population: Daily step counts were collected and reported for Secondary Outcome 12. Any reported falls were collected and reported as Adverse Events. Patient diaries were not collected, and no analysis was possible for other data recorded, such as daily activity.
Arm/Group | emPOWER Ankle (Powered Prosthesis)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of informed consent through study completion for each study subject, up to 12 months. All adverse events were monitored until they are adequately resolved, explained or the subject has exited the study.
Description: Definitions match clinicaltrials.gov
Groups:
- emPOWER Ankle (Powered Prosthesis): emPOWER Ankle: The device is 510k cleared and is intended to replace a missing foot and ankle. The emPOWER Ankle is to be used exclusively for fittings of lower-extremity amputations as prescribed by a healthcare professional.
  The subjects were fit with the emPOWER Ankle and followed for 3-4 months. After crossing over the passive foot and wearing it for 2 weeks, the subjects crossed over back to wearing the emPOWER Ankle up to the 12 months after the initial fitting.
- Subject's Own Passive Prosthesis: Subject's own passive prosthesis: Devices varied.
  The subject's own passive prosthesis was used as a baseline/control. No adverse events were collected prior to initial fitting with the emPOWER Ankle. After wearing the emPOWER Ankle for 3-4 months, subjects crossed over back to the passive prosthesis and wore it for 2 weeks. Subjects were crossed over back to the emPOWER for long-term follow up, up to 12 months after the initial fitting.
Arm/Group | emPOWER Ankle (Powered Prosthesis) | Subject's Own Passive Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/4
Other Adverse Events (participants affected / at risk) | 4/8 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | emPOWER Ankle (Powered Prosthesis) (N=8) | Subject's Own Passive Prosthesis (N=4)
Pancreatitis and ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0) — Subject was hospitalized due to vomiting approximately 6 weeks prior to the 6 Month Study Visit. He was admitted and diagnosed with pancreatitis and ketoacidosis.
Angioplasty (Cardiac disorders) | 1 (1) | 0 (0) — A subject reported having had an angioplasty procedure at the time of withdrawing consent. This event was not related to the device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | emPOWER Ankle (Powered Prosthesis) (N=8) | Subject's Own Passive Prosthesis (N=4)
Blisters (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Falls (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02958553/Prot_SAP_000.pdf